CLINICAL TRIAL: NCT03357198
Title: Correlation of Cough Peak Flow Measurement by an Electronic Handheld Spirometer Connected to the Endotracheal Tube and by the Intensive Care Unit Ventilator Flowmeter.
Brief Title: Correlation of Two Methods for Cough Peak Flow Measurement in Intubated Patients
Acronym: COUGH-ICU
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Other Study IDs: CHRO-2017-02
Record Dates: First submitted 2017-11-24; First posted 2017-11-29 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Respiratory Insufficiency; Ventilator Weaning
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cough peak flow measurement: All enrolled patients will undergo measurement of cough peak flow by two methods, i.e. using a handheld electronic spirometer, and using the ventilator flowmeter, in a randomized order.

SUMMARY:
Cough Peak Flow (CPF) seems to be an efficient tool to assess cough capacity for the intensive care unit (ICU) ventilated patient. CPF can be used in the ventilator weaning process, as reflecting the upper airways protection capacity.

CPF requires disconnection of the patient from the ICU ventilator, supplemental material (handheld spirometer, antibacterial filter) and an excellent synchronization between the specialized caregiver and the patient.

We aimed that CPF with the ventilator built-in flow-meter is correlated with CPF using a handheld flowmeter connected to the endotracheal tube.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Mechanically ventilated patient > 24 hours
* Weaning ventilator phase (PEEP < 9 cmH2O and Support < 15 cm H2O)
* Richmond Agitation Sedation Scale between -1 and +1
* Patient's agreement to participate

Exclusion Criteria:

* Pregnant women
* Bronchospasm
* FiO2 > 70%
* Thoracic surgery < 7 days
* Abdominal surgery < 7 days
* Thoracic injury with rib fracture < 21 days
* Pneumothorax < 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients undergoing invasive mechanical ventilation, sufficiently awake and cooperative to be assessed for their cough strength.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2018-08-29 (Actual); Study Completion 2018-08-29 (Actual)

PRIMARY OUTCOMES:
Correlation coefficient for the two CPF assessment methods, on extubation day | Within 1 hour before mechanical ventilation termination (extubation)
  Correlation coefficient for the two CPF assessment methods, on extubation day

SECONDARY OUTCOMES:
Discriminatory power of CPF to predict successful weaning of mechanical ventilation, i.e. no reintubation within 72 hours after extubation, or unsuccessful weaning. | During the mechanical ventilation until 72 hours post extubation
  Thresholds of CPF will be tested as predictors of weaning success
Assess the correlation between CPF and length of mechanical ventilation | During the mechanical ventilation until 72 hours post extubation
  Assess the correlation between CPF and length of mechanical ventilation
3. Correlation between the two CPF assessment methods the days before extubation | During the mechanical ventilation until 72 hours post extubation
  3. Correlation between the two CPF assessment methods the days before extubation

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume FOSSAT, Principal Investigator — CHR Orléans
Locations (1):
- CHR d'Orléans, Orléans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smina M, Salam A, Khamiees M, Gada P, Amoateng-Adjepong Y, Manthous CA. Cough peak flows and extubation outcomes. Chest. 2003 Jul;124(1):262-8. doi: 10.1378/chest.124.1.262. PMID 12853532
- [Background] Su WL, Chen YH, Chen CW, Yang SH, Su CL, Perng WC, Wu CP, Chen JH. Involuntary cough strength and extubation outcomes for patients in an ICU. Chest. 2010 Apr;137(4):777-82. doi: 10.1378/chest.07-2808. Epub 2010 Jan 22. PMID 20097804
- [Background] Macintyre NR. Evidence-based assessments in the ventilator discontinuation process. Respir Care. 2012 Oct;57(10):1611-8. doi: 10.4187/respcare.02055. PMID 23013898
- [Background] Thille AW, Richard JC, Brochard L. The decision to extubate in the intensive care unit. Am J Respir Crit Care Med. 2013 Jun 15;187(12):1294-302. doi: 10.1164/rccm.201208-1523CI. PMID 23641924